CLINICAL TRIAL: NCT01260493
Title: Continuum of Care, From the Emergency Ward to Living at Home - Implementation and Evaluation of an Intervention for Frail Elderly People
Brief Title: Continuum of Care for Frail Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vardalinstitutet The Swedish Institute for Health Sciences (Other)
Collaborators: VinnVård (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VårdkedjaVårdal
Record Dates: First submitted 2010-11-30; First posted 2010-12-15 (Estimated); Results first posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-06

CONDITIONS: Frail Elderly People
Keywords: very frail; case manager; integrated care; multiprofessional; intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional care, controlgroup (No Intervention): conventional care, control group
- integrated health care chain (Experimental): integrated health care chain. Geriatric assessment at emergency department (ED), case manager with multiprofessional team in the community, support for informal caregivers
  Interventions: Other: integrated health care chain

INTERVENTIONS:
Other: integrated health care chain — Geriatric assessment at ED, case manager with multiprofessional team in the community, support for informal caregivers
  Arms: integrated health care chain

SUMMARY:
The present study "Continuum of care for frail elderly people" form part of the research programme "Support for frail elderly persons - from prevention to palliation" (www.vardalinstitutet.net) which comprises research into three interventions. The program comprises interventions addressing frail elderly people in different phases of the disablement process, from elderly people who are beginning to develop frailty to very frail elderly people receiving palliative care.

The intervention "Continuum of care for frail elderly people" addresses elderly people who are frail and that have a great risk of high health care consumption. The hypothesis is that an intervention program for frail elderly people can reduce the number of visits to the emergency department, increase the life satisfaction and maintain the functional ability. The intervention, including an early geriatric assessment at the emergency department, early family support, a case manager in the community with a multi-professional team and active follow-up by the case manager, contributes to early recognition of the elderly people's need of information, care and rehabilitation and of informal caregivers' need of information. It enhances the transfer of information and integrates the care between different caregivers and different care levels, thereby better recognize frail elderly people's needs. Specifically, this study is expected to show that the intervention has a positive effect on the frail elderly person's functional ability, life satisfaction, satisfaction with health and social care, and health care consumption.

ELIGIBILITY:
Inclusion Criteria:

* 80 years and older or 65 to 79 years and having at least one chronic disease and being dependent in at least one activity of daily living

Exclusion Criteria:

* acute severely sick who immediately needs the assessment of a physician (within ten minutes)
* those with diagnosis of dementia (or severe cognitive impairment)
* patients in palliative care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 181 (Actual)
Dates: Start 2008-10; Primary Completion 2010-06 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Wilhelmson, MD,PhD, Principal Investigator — Göteborg University
Locations (1):
- University of Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Derived] Eklund K, Wilhelmson K, Gustafsson H, Landahl S, Dahlin-Ivanoff S. One-year outcome of frailty indicators and activities of daily living following the randomised controlled trial: "Continuum of care for frail older people". BMC Geriatr. 2013 Jul 22;13:76. doi: 10.1186/1471-2318-13-76. PMID 23875866
- [Derived] Hasson H, Blomberg S, Duner A. Fidelity and moderating factors in complex interventions: a case study of a continuum of care program for frail elderly people in health and social care. Implement Sci. 2012 Mar 22;7:23. doi: 10.1186/1748-5908-7-23. PMID 22436121
- [Derived] Wilhelmson K, Duner A, Eklund K, Gosman-Hedstrom G, Blomberg S, Hasson H, Gustafsson H, Landahl S, Dahlin-Ivanoff S. Design of a randomized controlled study of a multi-professional and multidimensional intervention targeting frail elderly people. BMC Geriatr. 2011 May 14;11:24. doi: 10.1186/1471-2318-11-24. PMID 21569570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recrutment period October 2008 to July 2011
Pre-assignment Details: exluded due to sheltered housing (n=2), dementia (n=1),palliative care (n=1) and died before baseline (n=4), declined particapation (n=12)
Groups:
- Integrated Health Care Chain: integrated health care chain. Geriatric assessment at emergency department (ED), case manager with multiprofessional team in the community, support for informal caregivers
  integrated health care chain : Geriatric assessment at ED, case manager with multiprofessional team in the community, support for informal caregivers
Period: Overall Study
Arm/Group | Conventional Care, Controlgroup | Integrated Health Care Chain
Started | 92 | 89
Completed | 76 | 85
Not Completed | 16 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Care, Controlgroup | Integrated Health Care Chain | Total
Number analyzed (Participants) | 76 | 85 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 76 | 85 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.1 (5.8) | 82.7 (5.2) | 82.4 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 47 | 89
  Male | 34 | 38 | 72
Region of Enrollment [Number; unit: participants]
  Sweden | 76 | 85 | 161

OUTCOME MEASURES:

1. Primary Outcome: Health Care Consumption
Description: Number of hospital days and admission will be analysed
Time Frame: 1 year
Reporting Status: Not Posted

2. Primary Outcome: Dependence in Activities of Daily Living
Description: Changes in number of person dependent in one or more daily activity from baseline to follow-up.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Conventional Care, Controlgroup | Integrated Health Care Chain
Number analyzed (Participants) | 76 | 85
participants | 18 | 33 [1.03 to 4.06]

3. Primary Outcome: Satisfaction With Health and Social Care
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Conventional Care, Controlgroup | Integrated Health Care Chain
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/85
Other Adverse Events (participants affected / at risk) | 0/76 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No